CLINICAL TRIAL: NCT00218257
Title: Interactions Between Progesterone and Cocaine in Women
Brief Title: Progesterone for the Treatment of Cocaine Dependence - 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 0205M23681; R01DA014573 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Results first posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Cocaine Abuse; Cocaine-Related Disorders
Keywords: Cocaine
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Progesterone

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive either progesterone or placebo during month 1, then crossover in month 2.
  During each month, participants will be randomized to receive either an active or inactive dose of cocaine during a 4-day in-hospital testing visit for a total of 4 testing days with self-administered cocaine.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Progesterone (Active Comparator): 200mg progesterone twice daily
  Interventions: Drug: Progesterone
- Placebo (Placebo Comparator): Placebo twice daily
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Progesterone — 200mg progesterone twice daily
  Other Names: prometrium
  Arms: Progesterone
Other: Placebo — placebo
  Arms: Placebo

SUMMARY:
Past research has demonstrated that cocaine dependent women experience less severe responses to cocaine during the luteal phase of the menstrual cycle, when estrogen and progesterone concentrations are high. The purpose of this study is to determine whether administered progesterone reduces subjective and physiological responses to cocaine in cocaine dependent individuals.

DETAILED DESCRIPTION:
Changes in ovarian hormones across the menstrual cycle impact responses to cocaine in women. Studies have shown that cocaine's effects are dampened during the luteal phase of the menstrual cycle, when estrogen and progesterone concentrations are high, relative to the other phases of the cycle, when concentrations of these hormones are relatively low. The purpose of this study is to determine whether progesterone reduces subjective and physiological responses to cocaine in cocaine dependent individuals. In addition, this study will help to advance the possibility of hormonal progesterone and pharmacologically-related drugs as potential treatment components for cocaine abuse.

Participants will undergo two 4-day inpatient periods, totaling 8 days of treatment. For women, the inpatient periods will occur during two consecutive menstrual cycles; for men, these will occur during two consecutive months. On Day 1, participants will receive a first dose of either progesterone or placebo. On Day 2, participants will receive a second and third dose of study medication. Participants will also participate in an adaptation session, which will familiarize the participant with the smoking equipment that will be used the following day. On Day 3, participants will receive a fourth dose of medication 2 hours prior to a smoking lab session. Prior to beginning the smoking lab session, participants will be asked to rate their current cocaine craving, anxiety level, appetite, and premenstrual symptoms. Participants will then be given a sample of the cocaine dose for the given day. During the smoking lab session, participants will be asked additional cocaine craving questions at pre-determined intervals and will be given the option to trade in previously earned tokens for either money or a dose of cocaine. Following completion of the smoking lab session, participants will receive their fifth dose of medication.

ELIGIBILITY:
Inclusion Criteria:

* Smoked at least 1 gram of cocaine each week for the 6 months prior to study entry
* Agrees to use an adequate method of contraception for the duration of the study
* If female, current regular menses

Exclusion Criteria:

* Major psychiatric illnesses, including psychotic mood and anxiety disorders
* Current dependence on alcohol or drugs other that cocaine or nicotine
* History of major medical illnesses, including liver disease, abnormal vaginal bleeding, suspected or known breast cancer, thrombophlebitis, or other medical conditions
* Current use of oral contraceptives or other types of hormonal contraceptives
* Amenorrhea
* Currently on parole or probation
* Received treatment for chemical dependency within the 6 months prior to study entry
* Known allergy to progesterone or peanuts

Ages: 18 Years to 46 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2002-07; Primary Completion 2008-04 (Actual); Study Completion 2008-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheila M. Specker, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 96 participants were consented. 45 participants began the first in-hospital study visit. The remaining 41 participants were lost to follow-up or chose not to participant after consenting. 45 participants completed the first 4-day inpatient study visit. 38 participants began and completed the second inpatient study visit.
Period: Intervention 1
Arm/Group | Progesterone, Then Placebo | Placebo, Then Progesterone
Started | 23 | 22
Completed | 23 | 22
Not Completed | 0 | 0
Period: Period Between Visit 1 and 2
Arm/Group | Progesterone, Then Placebo | Placebo, Then Progesterone
Started | 23 | 22
Completed | 19 | 19
Not Completed | 4 | 3
Not completed — Lost to Follow-up | 4 | 3
Period: Intervention 2
Arm/Group | Progesterone, Then Placebo | Placebo, Then Progesterone
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Cross-over design; All participants who completed baseline testing during study visit one are pooled and reported here.
Groups:
- All Participants: Cross-over design; all participants who completed the first of two inpatient study visits are pooled and reported here
Arm/Group | All Participants
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 45
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 25
  White | 12
  More than one race | 0
  Unknown or Not Reported | 7
Region of Enrollment [Number; unit: participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: Decision to Self-Administer Cocaine
Description: During 1 inpatient testing day, participants were given the opportunity to spend 5 earned tokens on either an active dose of cocaine or to keep the tokens for a $5 reward for each token. Decisions were solicited every 30 minutes. Outcome measure is reported as the percent of 5 decisions for which the participant chose to self-administer cocaine. 0% indicates that all 5 tokens were retained and traded for monetary reward. 100% indicates that the participant spent all 5 tokens on cocaine for self-administration.
  On another inpatient day, participants were offered the same 5 choices but with a inactive dose of cocaine (amount of cocaine insufficient for psychoactive effect) or a $5 monetary reward. 0% indicates that all 5 tokens were retained and traded for monetary reward. 100% indicates that the participant spent all 5 tokens on inactive doses of cocaine for self-administration.
  The order of days (active or inactive cocaine dosage) was random.
Time Frame: 4 days
Population: Only participants who completed both 4-day in-hospital testing visits are included in outcome measure reporting.
Measure: Mean (Standard Error); unit: percent of available doses
Groups:
- Progesterone: Progesterone (200mg, twice daily)
- Placebo: Placebo (given twice daily)
Arm/Group | Progesterone | Placebo
Number analyzed (Participants) | 38 | 38
percent of available doses
  Active Cocaine Dose | 66 (3.5) | 66 (3.3)
  Inactive Cocaine Dose | 32 (3.5) | 32 (3.3)

2. Secondary Outcome: Heart Rate
Description: During 1 inpatient testing day, participants were given the opportunity to spend 5 tokens on either an active dose of cocaine or to keep the tokens for a $5 reward each. Decisions were solicited every 30 minutes. There was a total of 5 decisions solicited. On another inpatient day, participants were offered the same 5 choices but with a inactive dose of cocaine or a monetary reward. The order of days (active or inactive cocaine dosage) was random. These 2 testing days were completed during a 4-day in-hospital testing session under the progesterone condition and placebo condition. Order of progesterone and placebo conditions were randomized.
  Heart rate was taken 2.5 minutes following administration of cocaine (active or inactive dosage). Up to 5 HR measurements were recorded based on participant decision to self-administer cocaine or not. Mean across up to 5 measures was calculated. Outcome is reported as the mean of mean measures during each of 4 study conditions.
Time Frame: 4 days
Population: Only participants who completed both 4-day in-hospital testing visits are included in outcome measure reporting.
Measure: Mean (Standard Deviation); unit: beats per minute
Groups:
- Progesterone: Progesterone (200mg, given twice daily)
Arm/Group | Progesterone | Placebo
Number analyzed (Participants) | 38 | 38
beats per minute
  Active Cocaine Dose | 87.9 (16.0) | 87.2 (16.3)
  Inactive Cocaine Dose | 77.6 (13.0) | 74.6 (12.1)

3. Secondary Outcome: Systolic Blood Pressure
Description: During 1 inpatient testing day, participants were given the opportunity to spend 5 tokens on either an active dose of cocaine or to keep the tokens for a $5 reward each. Decisions were solicited every 30 minutes. There was a total of 5 decisions solicited. On another inpatient day, participants were offered the same 5 choices but with a inactive dose of cocaine or a monetary reward. The order of days (active or inactive cocaine dosage) was random. These 2 testing days were completed during a 4-day in-hospital testing session under the progesterone condition and placebo condition. Progesterone and placebo conditions were randomized.
  Blood pressure was taken 2.5 minutes following administration of cocaine (active or inactive dosage). Up to 5 BP measurements were recorded based on participant decision to self-administer cocaine or not. Mean across up to 5 measures was calculated. Outcome is reported as the mean of mean measures during each of 4 study conditions.
Time Frame: 4 days
Population: Only participants who completed both 4-day in-hospital testing visits are included in outcome measure reporting.
Measure: Mean (Standard Deviation); unit: mmHG
Groups:
- Progesterone: Progesterone (200mg twice daily)
Arm/Group | Progesterone | Placebo
Number analyzed (Participants) | 38 | 38
mmHG
  Active Cocaine Dose | 129.9 (19.8) | 131.8 (18.5)
  Inactive Cocaine Dose | 117.4 (16.6) | 120.2 (17.6)

4. Secondary Outcome: Diastolic Blood Pressure
Description: as for outcome 3
Time Frame: 4 days
Population: Only participants who completed both 4-day in-hospital testing visits are included in outcome measure reporting.
Measure: Mean (Standard Deviation); unit: mmHG
Groups:
- Progesterone: Progesterone (200mg given twice daily)
Arm/Group | Progesterone | Placebo
Number analyzed (Participants) | 38 | 38
mmHG
  Active Cocaine Dose | 77.6 (12.6) | 78.6 (10.7)
  Inactive Cocaine Dose | 71.3 (8.8) | 72.2 (10.1)

5. Secondary Outcome: Cocaine Craving
Description: During 1 inpatient testing day, participants were given the opportunity to spend 5 tokens on either an active dose of cocaine or to keep the tokens for a $5 reward each. Decisions were solicited every 30 minutes. There was a total of 5 decisions solicited. On another inpatient day, participants were offered the same 5 choices but with a inactive dose of cocaine or a monetary reward. The order of days (active or inactive cocaine dosage) was random. These 2 testing days were completed during a 5-day in-hospital testing session under the progesterone condition and placebo condition. Progesterone and placebo conditions were randomized.
  Participants were asked to rate cocaine craving on a scale of 0-5 prior to administration of cocaine (active or inactive dose). Lower scores indicate less cocaine craving.
Time Frame: 4 days
Population: Only participants who completed both 4-day in-hospital testing visits are included in outcome measure reporting.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Progesterone | Placebo
Number analyzed (Participants) | 38 | 38
score on a scale
  Active Cocaine Dose | 3.99 (.17) | 4.02 (.16)
  Inactive Cocaine Dose | 2.06 (.16) | 1.38 (.17)

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Progesterone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 1/38 | 0/38
Other Adverse Events (participants affected / at risk) | 14/38 | 0/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Progesterone (N=38) | Placebo (N=38)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Progesterone (N=38) | Placebo (N=38)
Headache (Nervous system disorders) | 7 | 0 (0)
GI Upset (Gastrointestinal disorders) | 7 (7) | 0 (0) — Nausea, vomiting, and diarrhea

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes